CLINICAL TRIAL: NCT00534482
Title: The Impact of Brief Primary Care Counseling and Novel Physiological Measures on Patient Physical and Emotional Health
Brief Title: Evaluation of the "Americans in Motion - Healthy Interventions" Project
Acronym: AIM-HI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Academy of Family Physicians (Other)
Collaborators: The PepsiCo Foundation (Other)
Responsible Party: Wilson Pace, MD, FAAFP, American Academy of Family Physicians; University of CO - Health Sciences
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 07-034
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Physical Activity; Diet; Mental Health
Keywords: fitness
MeSH Terms: conditions — Motor Activity; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A, 1, I (Experimental): Practice-level treatment group
  Interventions: Behavioral: Enhanced Office
- A, 1, II (Active Comparator): Practice-level comparison group
  Interventions: Behavioral: Conventional Office
- B, 1, I (Experimental): Patient-level treatment group
  Interventions: Behavioral: AIM-HI program with enhanced feedback
- B, 1, II (Active Comparator): Patient-level comparison group
  Interventions: Behavioral: AIM-HI program and regular feedback

INTERVENTIONS:
Behavioral: Enhanced Office — Clinicians and office staff personally engage in AIM-HI fitness program, and promote program to patients
  Arms: A, 1, I
Behavioral: Conventional Office — Conventional office: Clinicians and office staff are not personally engaged in the AIM-HI fitness program, but promote program to patients.
  Arms: A, 1, II
Behavioral: AIM-HI program with enhanced feedback — Patient receives feedback on two novel indicators of their individual cardiovascular risk that: 1)appear to relate to obesity and lack of physical activity, and 2) may show relatively rapid change with improvements in these areas. These are the Homeostatic Assay - Insulin Resistance or HOMA-IR and Nuclear Molecular Resonance (NMR) lipoprotein profiles (NMRLP). These patients and their physicians also will receive periodic feedback on other outcome measures, including BMI, blood pressure, a 3-minute step test, eating assessment, physical activity assessment, and emotional well-being assessment.
  Arms: B, 1, I
Behavioral: AIM-HI program and regular feedback — Patients will not receive feedback on two specific cardiovascular risk indicators (ie, Homeostatic Assay - Insulin Resistance, Nuclear Molecular Resonance lipoprotein profiles). However, patients will receive feedback on Body Mass Index, blood pressure, a 3-minute step test, eating assessment, physical activity assessment, and emotional well-being assessment.
  Arms: B, 1, II

SUMMARY:
This research project brings together the American Academy of Family Physicians (AAFP) National Research Network (AAFP-NRN) and the AAFP's public health initiative, Americans In Motion (AIM). This project will develop and evaluate a practice improvement program to improve family physicians' delivery of effective patient-centered behavior change interventions for "fitness" (physical activity, nutrition and emotional well-being). The investigators seek to develop a unique program that positions fitness in a central role as "the treatment of choice" when dealing with issues of prevention and treatment of chronic conditions. In addition, this newly developed program is intended to help shift the paradigm of family physicians' use of common advice-giving methods to more effective patient-centered lifestyle counseling. Ultimately, this program will seek to improve care for all patients through fitness-related physician interventions.

Outcomes: This study design will allow the investigators to evaluate whether (and how) dissemination of educational materials impacts patient intervention by first engaging clinicians and staff in their personal use of these materials. This project will also evaluate the effects of the behavioral change tools, as well as, the added impact of new physiologic feedback measures (HOMA-IR and NMR Lipoprotein profiles) on physical activity and diet in study participants.

Conclusion: Primary care offices can become more effective settings to help patients improve physical activity, diet and emotional well-being. Demonstrating the value and impact of creating "healthy offices" that endorse and support clinicians, office staff and patients in the use of effective educational materials fits well with the new model of care as part of the AAFP's "Future of Family Medicine" initiatives, which emphasize the importance of lifestyle decisions and supporting successful changes in behaviors within primary care. This project will help define how to accomplish this.

DETAILED DESCRIPTION:
Study Design: This trial will consist of a two-level randomized controlled trial. The first level of randomization will be performed at the practice level in order to study the impact of involving both clinicians and office staff in making their own personal changes (i.e., creating the "healthy" office)- a central component of AIM - on the translation of the project's educational tools to patients. The second level of randomization will occur at the patient level comparing two practice level interventions designed to improve nutrition, increase physical activity and improve emotional well-being. Furthermore, the effectiveness of the educational tools will be evaluated on self-reported diet, physical activity and emotional well-being and established physiologic measures on behavioral change. Both arms of the study will receive brief office-based counseling using established tools that have been compiled for this project. Practices will be asked to work on incorporating brief nutrition, physical activity and emotional well-being messages into routine care - either motivational in nature for people not willing to work on lifestyle changes, or goal-oriented for those working on changes. Patients in the intervention arm will also receive feedback concerning changes in two novel physiologic measures that correlate with improved nutrition and increased physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* BMI greater than or equal to 30
* Able to participate in moderate physical activity including a 3-minute step test without worsening an existing medical condition
* Life expectancy of greater than one year
* Able to read English or Spanish; and
* Able to be contacted via phone for follow-up with project staff

Exclusion Criteria:

* Too ill to participate
* A current diagnosis at the index visit of type 2 diabetes, hyperlipidemia, or coronary heart disease
* Doctor's evaluation of patient as not appropriate for physical activity
* Not capable of giving informed consent; and
* Unable to read English or Spanish, including blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Aggregate patient assessment of practice involvement in patient health behaviors | 12 months
Aggregate clinician and practice staff assessment of practice involvement in patient healthy behaviors | 12 months
Spread of billing codes for physician fitness counseling | 12 months
Body Mass Index | baseline, 6, 9, and 12 months
Homeostatic Assay- Insulin Resistance | baseline, 3, 6, 9, and 12 months
Nuclear Molecular Resonance (NMR) Lipoprotein Profiles | baseline, 3, 6, 9, and 12 months
3-Minute Step Test | baseline, 3, 6, 9, and 12 months
Blood Pressure | baseline, 3, 6, 9, and 12 months

SECONDARY OUTCOMES:
Functional health status | baseline, 3, 6, 9, and 12 months
Quality of life and well-being | baseline, 3, 6, 9, and 12 months
Treatment self-regulation items related to diet | baseline, 3, 6, 9, and 12 months
Treatment self-regulation items related to physical activity | baseline, 3, 6, 9, and 12 months
Perceived competence for maintaining healthy eating | baseline, 3, 6, 9, and 12 months
Perceived competence for maintaining physical activity | baseline, 3, 6, 9, and 12 months
Perceived competence for maintaining emotional health | baseline, 3, 6, 9, and 12 months
Diet and nutrition related items | baseline, 3, 6, 9, and 12 months
Physical activity related items | baseline, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wilson D Pace, MD, FAAFP, Principal Investigator — American Academy of Family Physicians
Locations (1):
- American Academy of Family Physicians National Research Network, Leawood, Kansas, United States

REFERENCES:
- [Background] Stern SE, Williams K, Ferrannini E, DeFronzo RA, Bogardus C, Stern MP. Identification of individuals with insulin resistance using routine clinical measurements. Diabetes. 2005 Feb;54(2):333-9. doi: 10.2337/diabetes.54.2.333. PMID 15677489
- [Background] Shadid S, LaForge R, Otvos JD, Jensen MD. Treatment of obesity with diet/exercise versus pioglitazone has distinct effects on lipoprotein particle size. Atherosclerosis. 2006 Oct;188(2):370-6. doi: 10.1016/j.atherosclerosis.2005.10.038. Epub 2005 Nov 28. PMID 16313908
- [Background] McClernon FJ, Yancy WS Jr, Eberstein JA, Atkins RC, Westman EC. The effects of a low-carbohydrate ketogenic diet and a low-fat diet on mood, hunger, and other self-reported symptoms. Obesity (Silver Spring). 2007 Jan;15(1):182-7. doi: 10.1038/oby.2007.516. PMID 17228046